CLINICAL TRIAL: NCT07375459
Title: Mobile-assisted Brief Intervention for Smoking Cessation in Community-based Setting: a Pilot Randomised Controlled Trial
Brief Title: Community-based Mobile-assisted Brief Intervention for Smoking Cessation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, LUK Tzu Tsun, Assistant Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NUS-IRB-2025-690
Record Dates: First submitted 2026-01-22; First posted 2026-01-29 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Smoking &Amp; Tobacco Cessation
Keywords: mHealth; WhatsApp; smoking cessation; chat-based intervention; Singapore
MeSH Terms: conditions — Smoking; Tobacco Use Cessation; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile-assisted brief intervention (Experimental)
  Interventions: Behavioral: Brief cessation advice + self-help booklet; Behavioral: Opt-out referral; Behavioral: Mobile chat messaging
- Brief advice (Active Comparator)
  Interventions: Behavioral: Brief cessation advice + self-help booklet

INTERVENTIONS:
Behavioral: Brief cessation advice + self-help booklet — Participants will receive brief cessation advice following the AWARD (ask, warn, advise, refer, do-it-again) model and a 24-page self-help booklet.
Behavioral: Opt-out referral — Research personnel will assist the participant in signing up for the I Quit Programme to receive additional cessation support, unless they decline
  Arms: Mobile-assisted brief intervention
Behavioral: Mobile chat messaging — Participants will receive personalised chat-based support delivered by a live counsellor for 3 months via WhatsApp. The message will incorporate behaviour change techniques for smoking cessation and mindfulness principles to strengthen participants' capacity to quit smoking.
  Arms: Mobile-assisted brief intervention

SUMMARY:
The goal of this pilot trial is to evaluate the feasibility of a mobile-assisted brief intervention for smoking cessation in community-based individuals in Singapore. Specific aims include:

1. To assess how many eligible individuals accept the invitation to participate in the trial
2. To assess the retention of the participants through 6 months after treatment initiation
3. To assess the acceptability of the intervention in terms of participants' engagement and ratings
4. To examine the intervention effect on abstinence outcomes

Participants will be randomly assigned to either the intervention group or control group and followed for 6 months from randomisation.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21 to 80 years
* Smoked at least one cigarette daily
* Able to communicate and read in English or Chinese
* Own a smartphone with WhatsApp installed

Exclusion Criteria:

* Exposed to any smoking cessation treatment in the past 3 months
* Pregnant women

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Biochemically validated smoking abstinence rate | 6 months
  Defined as an exhaled carbon monoxide level of <5 parts per million or a negative salivary cotinine test (cut off 30ng/mL)
Recruitment rate | 6 months
  Number of participants divided by the number of eligible subjects
Retention rate | 6 months
  Number of participants completed the follow-up divided by the number of participants

SECONDARY OUTCOMES:
Self-reported 7-day point-prevalence smoking abstinence rate | 3 months
  Being completely smoke-free in the past 7 days
Self-reported 7-day point-prevalence smoking abstinence rate | 6 months
  Being completely smoke-free in the past 7 days
Self-reported smoking reduction rate | 3 months
  Smoking reduction by at least half of the baseline daily number of cigarettes in individuals who continue to smoke
Self-reported smoking reduction rate | 6 months
  Smoking reduction by at least half of the baseline daily number of cigarettes in individuals who continue to smoke
Self-reported quit attempt rate | 3 months
  Serious quit attempt that lasted 24 hours or longer
Self-reported quit attempt rate | 6 months
  Serious quit attempt that lasted 24 hours or longer
Smoking cessation service use rate | 3 months
  Use of any smoking cessation service during the follow-up period
Smoking cessation service use rate | 6 months
  Use of any smoking cessation service during the follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Tzu Tsun Luk, PhD, RN, Principal Investigator — National University of Singapore
Locations (1):
- National University of Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No